CLINICAL TRIAL: NCT00831636
Title: A Phase I/II Study of CP-4055 in Patients With Platinum Resistant Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clavis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP4055-204
Record Dates: First submitted 2009-01-28; First posted 2009-01-29 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Ovarian Cancer
Keywords: CP-4055; Cancer; Metastatic; Solid tumors; advanced ovarian cancer; stage III and IV ovarian cancer; advanced epithelian ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — 5'-oleoyl cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label CP-4055 (Experimental): Phase I: Dose escalation Phase II: Fixed dose
  Interventions: Drug: CP-4055

INTERVENTIONS:
Drug: CP-4055 — D1-5 and D8(+2)-12(+2) q4w
Drug: CP-4055 — IV administration day 1-5 and day 8-12 in a 4 week schedule

SUMMARY:
This is non randomised, open label, dose finding, efficacy and safety study, enrolling patients with advanced (stage III and IV) ovarian cancer It will be conducted in two successive phases. Phase II has a two-step design

DETAILED DESCRIPTION:
Phase I

* Three eligible patients will be enrolled at each dose level (DL), according to standard dose escalation decision rules
* Patients will receive CP-4055 at increasing DLs until the maximum tolerated dose and the recommended dose (RD) have been established

Phase II

* Step 1 (The patient inclusion may stop after this step):

  * Patients will be enrolled at the RD until there are maximum 16 evaluable patients at this DL
* Step 2:

  * Depending on the response rate at step 1, up to 26 patients will be included and treated at step 2

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented advanced epithelial ovarian cancer measurable with CT and/or MRI
* Received prior chemotherapy regimen(s) for ovarian cancer, at least one being a platinum based therapy (PBT)
* Evidence of platinum resistant or refractory disease
* ECOG Performance Status 0 - 1
* Life expectancy > 3 months
* Signed informed consent (IC)
* Women of child-bearing potential must have a negative serum or urine pregnancy test. Nursing patients are excluded.
* Women of child-bearing potential must not become pregnant while participating in the study
* Adequate haematological and biological functions

Exclusion Criteria:

* Patients with mixed mullerian tumours (MMT) (carcinosarcomas)
* Known brain metastases
* Another known active cancer within the last 5 years
* Radiotherapy to more than 30 % of bone marrow
* Participation in another therapeutic clinical study within 30 days of enrolment or during this clinical study
* Concomitant treatment with a non-permitted medication
* A history of allergic reactions or sensitivity attributed to compounds of similar or biological composition to CP-4055, i.e., ara-C and/or egg
* Any serious concomitant systemic disorders incompatible with the clinical study
* Any significant CNS or psychiatric disorder(s) that would hamper the patient's compliance
* Pregnancy or breastfeeding
* Known positive status for HIV and/or hepatitis B or C
* Drug and/or alcohol abuse
* Any reason why, in the investigator's opinion, the patient should not participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Phase I: Determine recommended dose for phase II studies of CP-4055 when given five consecutive days twice in a 4 week schedule, D1-5 and D8(+2)-12(+2) q4w | August 2009/June 2010
Phase II: Determine the antitumour activity of CP-4055 | August 2009/June 2010

SECONDARY OUTCOMES:
Determine pharmacokinetic (PK) parameters | August 2009/June 2010
Explore the time to progression (TTP) | August 2009/June 2010
Investigate the duration of tumour response | August 2009/June 2010
Determine the nature and degree of toxicity of CP-4055 in this patient population | August 2009/June 2010

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, MD, Principal Investigator — Medical Oncology B, National Cancer Institute, Via Mariano Semmola, IT-80131 Naples, Italy
Locations (5):
- U.Z. Gasthuisberg, Gynecologic Oncology, Herestraat 49, Leuven, Belgium
- Italy (4):
  - Medical Oncology C, National Cancer Institute, Centro di Riferimento Oncologico, Aviano (PN)
  - Medical Oncology B, National Cancer Institute, Via Mariano Semmola, Naples
  - Department of Oncology, Catholic University of the Sacred Heart, Rome
  - Medical Oncology, Fatebenefratelli Hospital, Isola Tiberina, Rome

REFERENCES:
- See also: Clavis Pharma Home Page — http://www.clavispharma.com/